CLINICAL TRIAL: NCT05320393
Title: Phase II Multi-Ctr, Prospective, Randomized, Double Blind, Active-Controlled Single Treatment Increasing Dose Trial to Study Safety & Duration of Effect of 40U of PrabotulinumtoxinA-xvfs in Adult Subjects for Treatment of Glabellar Lines
Brief Title: Study to Demonstrate Safety and Duration of Effect of 40 Units of PrabotulinumtoxinA-xvfs to Treat Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evolus, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVOLUS-CLIN201
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-06

CONDITIONS: Glabellar Frown Lines
Keywords: Botulinum toxin type A
MeSH Terms: interventions — prabotulinumtoxin A; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug (Experimental): 40U of PrabotulinumtoxinA-xvfs
  Interventions: Drug: PrabotulinumtoxinA-Xvfs
- OnabotulinumtoxinA (Active Comparator): 20U of OnabotulinumtoxinA
  Interventions: Drug: OnabotulinumtoxinA
- PrabotulinumtoxinA-xvfs (Active Comparator): 20U of PrabotulinumtoxinA-xvfs
  Interventions: Drug: PrabotulinumtoxinA-Xvfs

INTERVENTIONS:
Drug: PrabotulinumtoxinA-Xvfs — One treatment of 40 units
  Other Names: Jeuveau
  Arms: Study Drug
Drug: OnabotulinumtoxinA — One treatment of 20 units
  Other Names: Botox Cosmetic
  Arms: OnabotulinumtoxinA
Drug: PrabotulinumtoxinA-Xvfs — One treatment of 20 units
  Other Names: Jeuveau
  Arms: PrabotulinumtoxinA-xvfs

SUMMARY:
The purpose of this study is to demonstrate the safety and duration of effect of 40 Units of prabotulinumtoxinA-xvfs (Jeuveau®) in providing temporary improvement in the appearance of moderate to severe glabellar lines (frown lines, which are the vertical lines that develop between the eyebrows) in adult participants. It will also determine if the duration of effect of 40 Units of Jeuveau® is greater than that of 20 Units of Jeuveau® and 20 Units of Botox® Cosmetic.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind, active-controlled, single-treatment, increasing dose design. Up to one hundred and fifty subjects will be randomized 1:1:1, to either 20 Units onabotulinumtoxinA (Botox® Cosmetic), 20 Units prabotulinumtoxinA-xvfs (Jeuveau®), or 40 Units prabotulinumtoxinA-xvfs (Jeuveau®).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female of any race, 18 years of age or older.
* Female subjects of childbearing potential must have a negative urine pregnancy test during Visits 1 (Screening) and Visit 2 (if applicable) and practice a reliable method of contraception for the duration of the study.
* Moderate to severe glabellar lines (i.e., score of 2 or 3) on maximum frown as assessed by the investigator using the Glabellar Line Scale (GLS).
* Subject has moderate to severe glabellar lines (i.e., score of 2 or 3) at maximum frown as assessed by the subject using the GLS.
* Able to follow study instructions and likely to complete all required visits.
* Sign the Institutional Review Board (IRB) -approved Informed Consent Form (ICF) prior to any study-related procedures being performed.

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
* Known hypersensitivity or previous allergic reaction to any constituent of the Investigational Product (IP) or control.
* Any active infection in the area of the injection sites.
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart.
* Marked facial asymmetry (Investigator discretion).
* Ptosis of eyelid and/or eyebrow, or history of eyelid and/or eyebrow ptosis.
* History of facial nerve palsy.
* Excessive dermatochalasis, deep dermal scarring, thick sebaceous skin (Investigator discretion).
* Medical condition that may affect neuromuscular function (e.g., myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis).
* Previous treatment with botulinum toxin of any serotype above the level of the lateral canthus within the last 6 months.
* Planned treatment with botulinum toxin of any serotype below the level of the lateral canthus during the study period.
* Previous treatment with any facial aesthetic procedure (e.g., injection with biodegradable fillers, chemical peeling, photo rejuvenation) in the glabellar area within the last 12 months.
* Previous insertion of permanent material in the glabellar area.
* Any previous energy based or cryotherapy-based treatment of facial muscles superior to the lateral canthus.
* Any other planned facial aesthetic procedure during the trial period, superior to the level of the lateral canthus (can continue with their usual skin care routine).
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles, or a combination of these, or scars in the glabellar area and the surrounding areas (including eyebrow).
* Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
* Evidence of recent alcohol or drug abuse (Investigator discretion).
* History of poor cooperation or unreliability.
* Planning to move out of the area prior to study completion.
* Subjects who are investigational site staff members or family members of such employees.
* Exposure to any other investigational drug/device within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Avelar, MD, Study Director — Evolus, Inc.
Locations (1):
- Aesthetic Eyelid Plastic Surgery, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Drug | OnabotulinumtoxinA | PrabotulinumtoxinA-xvfs
Started | 51 | 50 | 53
Completed | 49 | 48 | 47
Not Completed | 2 | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Moved; too much driving | 0 | 0 | 2
Not completed — Did not receive treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug | OnabotulinumtoxinA | PrabotulinumtoxinA-xvfs | Total
Number analyzed (Participants) | 51 | 50 | 53 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.3) | 47.0 (11.1) | 46.8 (12.9) | 47 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 47 | 50 | 145
  Male | 3 | 3 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 15 | 51
  Not Hispanic or Latino | 31 | 34 | 37 | 102
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 48 | 47 | 49 | 144
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 53 | 154
Participant Has a Prior history of botulinum toxin use [Count of Participants; unit: Participants] — Participants were asked if they had ever been treated with botulinum toxin for any indication and participants responded yes or no
  Participants | 26 | 26 | 19 | 71
Glabellar Line Score of Moderate at Maximum Frown by Investigator Assessment [Count of Participants; unit: Participants] — Validated 4-point Glabellar Line Scale (GLS): 0=None/No lines, 1=Mild/Line seen, not sharp, 2=Moderate/Line sharper, deep, may see heaping of skin; 3=Severe/Deeper line, heaping of skin, skin may be opposed
  Participants | 15 | 14 | 18 | 47
Glabellar Line Score of Moderate at Maximum Frown by Subject Assessment [Count of Participants; unit: Participants] — Validated 4-point Glabellar Line Scale (GLS): 0=None/No lines, 1=Mild/Line seen, not sharp, 2=Moderate/Line sharper, deep, may see heaping of skin; 3=Severe/Deeper line, heaping of skin, skin may be opposed
  Participants | 11 | 7 | 13 | 31
Glabellar Line Score of Severe at Maximum Frown by Investigator Assessment [Count of Participants; unit: Participants] — VValidated 4-point Glabellar Line Scale (GLS): 0=None/No lines, 1=Mild/Line seen, not sharp, 2=Moderate/Line sharper, deep, may see heaping of skin; 3=Severe/Deeper line, heaping of skin, skin may be opposed
  Participants | 36 | 36 | 35 | 107
Glabellar Line Score of Severe at Maximum Frown by Subject Assessment [Count of Participants; unit: Participants] — Validated 4-point Glabellar Line Scale (GLS): 0=None/No lines, 1=Mild/Line seen, not sharp, 2=Moderate/Line sharper, deep, may see heaping of skin; 3=Severe/Deeper line, heaping of skin, skin may be opposed
  Participants | 40 | 43 | 40 | 123

OUTCOME MEASURES:

1. Primary Outcome: Duration of Effect Described by Kaplan-Meier Analysis
Description: Effectiveness of prabotulinumtoxinA 40 Units compared to prabotulinumtoxinA 20 Units will be assessed for each subject based on the number of days from baseline to the day that the Glabellar Line Scale (GLS) severity, by Investigator Assessment, returns to the baseline value. The treatment will be considered to remain effective for the amount of time during which the GLS severity at maximum frown has not returned to baseline severity.
Time Frame: Duration of effect for each subject will be based on number of days from baseline to the day that Glabellar Line Scale severity (Investigator Assessment) returns to baseline value, assessed every 30 days up to 365 days.
Population: 152 participants comprised the modified intent to treat population; all 152 participants had at least one post-treatment assessment for the primary efficacy endpoint.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Study Drug | OnabotulinumtoxinA | PrabotulinumtoxinA-xvfs
Number analyzed (Participants) | 51 | 50 | 51
Days | 183 [153 to 211] | 148 [121 to 174] | 149 [130 to 174]
Statistical Analysis 1: Comparison: Study Drug vs OnabotulinumtoxinA vs PrabotulinumtoxinA-xvfs; The primary effectiveness endpoint was a measure of duration of effect, described by Kaplan-Meier curves and the median times, with associated 2-sided 95% confidence intervals for each treatment group; Test type: Other — This study was not powered for formal hypothesis testing; analyses were intended for interpretation purposes only. Analysis was performed using the modified Intent-to-Treat population and regardless of responder status; p = 0.0109, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of up 12 months post treatment.
Description: Adverse events regardless of relationship or seriousness were collected at all study visits from the time of study enrollment until the follow-up or early termination visit period, and could be reported in response to a query, observed by the Investigator or site personnel, or reported spontaneously by the study participant.
Arm/Group | Study Drug | OnabotulinumtoxinA | PrabotulinumtoxinA-xvfs
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 2/51 | 5/50 | 3/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=51) | OnabotulinumtoxinA (N=50) | PrabotulinumtoxinA-xvfs (N=52)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the Study Sponsor. Any Investigator involved with this study is obligated to provide the Sponsor with complete test results and all data derived from the study.

DOCUMENTS (2):
  • Study Protocol (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT05320393/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT05320393/SAP_001.pdf